CLINICAL TRIAL: NCT00771433
Title: Evaluation of the Efficacy of Adding Daily G-CSF (Granulocyte Colony Stimulating Factor) for Prevention of Hematologic Toxicity Due to Neoadjuvant or Adjvuant Chemotherapy in Breast Cancer
Brief Title: G-CSF in Preventing Neutropenia in Women Receiving Chemotherapy for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000599535; FRE-CFB-LENO-SEIN; INCA-RECF0516; EUDRACT-2007-002753-23; FRE-CFB-CFB/2007-01; CHUGAI-FRE-CFB-LENO-SEIN
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2008-12

CONDITIONS: Breast Cancer; Chemotherapeutic Agent Toxicity; Neutropenia
Keywords: neutropenia; chemotherapeutic agent toxicity; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — Filgrastim

ARMS (2):
- Group 1 (Experimental): Patients receive filgrastim (G-CSF) subcutaneously (SC) once daily on days 6-11 of each course of chemotherapy as primary prophylaxis. Chemotherapy courses repeat every three weeks for 3-6 courses.
  Interventions: Biological: filgrastim
- Group 2 (Experimental): Patients receive G-CSF SC once daily on days 6-11 of each course of chemotherapy as primary prophylaxis. Chemotherapy courses repeat every three weeks for 3-6 courses. Patients may also receive secondary prophylaxis with G-CSF if they experience an episode of neutropenia.
  Interventions: Biological: filgrastim

INTERVENTIONS:
Biological: filgrastim — Given subcutaneously

SUMMARY:
RATIONALE: G-CSF may prevent or reduce febrile neutropenia in women receiving chemotherapy for breast cancer. It is not yet known which G-CSF regimen is more effective in preventing neutropenia.

PURPOSE: This phase II trial is studying how well G-CSF works in preventing neutropenia in women receiving chemotherapy for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of filgrastim (G-CSF) in preventing hematological toxicity in women with breast cancer receiving neoadjuvant or adjuvant chemotherapy.

Secondary

* Compare actual vs theoretical dose intensity.

OUTLINE: This is a multicenter study. Patients are stratified according to age (< 65 years vs ≥ 65 years) and prior chemotherapy (adjuvant vs neoadjuvant). Patients are assigned to 1 of 2 groups.

* Group 1: Patients receive filgrastim (G-CSF) subcutaneously (SC) once daily on days 6-11 of each course of chemotherapy as primary prophylaxis. Chemotherapy courses repeat every three weeks for 3-6 courses.
* Group 2: Patients receive G-CSF SC once daily on days 6-11 of each course of chemotherapy as primary prophylaxis. Chemotherapy courses repeat every three weeks for 3-6 courses. Patients may also receive secondary prophylaxis with G-CSF if they experience an episode of neutropenia.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer
* Receiving 1 of the following neoadjuvant or adjuvant chemotherapy regimens:

  * Six courses of epirubicin hydrochloride and docetaxel
  * Six courses of fluorouracil, epirubicin hydrochloride, and cyclophosphamide (FEC) 100 or 3 courses of FEC 100 and 3 courses of docetaxel 100
* Must have received at least 2 chemotherapy regimens prior to study therapy
* No malignant hematological disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No contraindications to standard neoadjuvant or adjuvant chemotherapy
* No known hypersensitivity to G-CSF or any of its components
* No patients deprived of liberty or under guardianship
* No psychological, familial, social, or geographical reasons preventing follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent participation in another experimental drug study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of febrile neutropenia

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Delcambre, Study Chair — Centre Francois Baclesse
Locations (1):
- Centre Regional Francois Baclesse, Caen, France